CLINICAL TRIAL: NCT01636791
Title: Cognitive Behavior Therapy Versus a Return to Work Intervention for Sick-listed Patients With Common Mental Illness in Primary Care: a Randomized Clinical Trial
Brief Title: CBT Versus a Return to Work Intervention for Patients With Common Mental Illness in Primary Care
Acronym: CBT vs RTW I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Hedman, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GVC CBT vs RTW
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Anxiety Disorders; Major Depression; Stress Disorders; Primary Insomnia
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder, Major; Stress Disorders, Traumatic; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Return to Work

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Behavior Therapy (Active Comparator): As the trial will include several different common mental disorders, the cognitive behavior therapy used in the study will be based on the protocols with best empirical support. Cognitive behavior therapy entails psychoeducational components, i.e. the patient is learns about the disorder and how to view it from a cognitive behavioral perspective. The most important part of the treatment is systematic behavior changes often targeted at exposure to feared stimuli. This is combined with cognitive interventions targeted at challenging negative automatic thoughts. All treatments will be delivered by licensed psychologists.
  Interventions: Behavioral: Cognitive behavior therapy
- Return to work (Experimental): Participants randomized to this arm will receive an experimental treatment, based in cognitive behavioral therapy, with primary aim to help patients return to work. Interventions are aimed at solving work-related problems and comprises problem-solving training and systematic employer-patient meetings aimed at facilitating a gradual return to the workplace. Licensed psychologists deliver all treatments.
  Interventions: Behavioral: Return to work
- CBT and Return to work (Experimental): Participants randomized to this arm will receive a combination of cognitive behavior therapy and the return to work treatment. This arm is included in the study as the clinically most relevant therapy, would the return to work treatment be effective in reducing sick leave, is a treatment were patients are provided support to return to work but also is clinically effective in reducing psychiatric symptoms.
  Interventions: Behavioral: Cognitive behavior therapy; Behavioral: Return to work

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Cognitive behavior therapy entails psychoeducational components, i.e. the patient is learns about the disorder and how to view it from a cognitive behavioral perspective. The most important part of the treatment is systematic behavior changes often targeted at exposure to feared stimuli. This is combined with cognitive interventions targeted at challenging negative automatic thoughts. All treatments will be delivered by licensed psychologists.
  Arms: CBT and Return to work; Cognitive Behavior Therapy
Behavioral: Return to work — Participants randomized to this arm will receive an experimental treatment, based in cognitive behavioral therapy, with primary aim to help patients return to work. Interventions are aimed at solving work-related problems and comprises problem-solving training and systematic employer-patient meetings aimed at facilitating a gradual return to the workplace. Licensed psychologists deliver all treatments.
  Arms: CBT and Return to work; Return to work

SUMMARY:
Background: Common mental illness, such as anxiety disorders and depression, is the main cause for sick leave in Sweden. Cognitive behavior therapy (CBT) has been shown to be effective in alleviating target symptoms of these disorders, but its effect on sick leave rates has not been sufficiently addressed. The investigators have developed an intervention called return to work (RTW), which is based in cognitive behavioral theory, that has a primary aim of helping sick-listed patients with common mental illness return to work. This new treatment has not been evaluated in a randomized controlled trial.

Aims: The aim of this study is to investigate the effect of CBT and RTW for common mental illness in a randomized controlled trial conducted in primary care. Participants will be randomized to diagnosis specific CBT (n=70), RTW (n=70), or a combination of the two treatments (n=70). Main outcomes are days of sick leave and clinician severity rating of psychiatric symptoms. This study could contribute to new knowledge regarding how to best treat patients on sick leave with common mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Have been on sick leave (at least 50%) for at least 1 month and not more than 6 months
* Have an anxiety disorder diagnosis (obsessive compulsive disorder, social phobia, panic disorder, generalized anxiety disorder, post-traumatic stress disorder, specific phobia), or/and major depression, or/and maladaptive stress reaction, or/and primary insomnia

Exclusion Criteria:

* A lower score than 4 on the Clinician severity rating scale
* A higher score than 6 on the Clinician severity rating scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sick leave | 1 year
  Number of days on sick leave
Clinician Severity Rating (CSR) | Baseine, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in CSR at post-treatment, 26 week follow-up, and 52 week follow-up compared to baseline.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale-Self-report (MADRS-S) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in MADRS-S at post-treatment, 26 week follow-up, and 52 week follow-up
Work ability index (WAI) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in WAI at post-treatment, 26 week follow-up, 52 week follow-up
Insomnia Severity Index (ISI) | Baseline, post-treatment (variable depending on disorder, 26 week follow-up, 52 week follow-up
  Change in ISI at post-treatment, 26 week follow-up, and 52 week follow-up
Health Anxiety Inventory (HAI) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in HAI at post-treatment, 26 week follow-up, and 52 week follow-up
Perceived Stress Scale (PSS) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in PSS at post-treatment, 26 week follow-up, and 52 week follow-up
Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in TIC-P at post-treatment, 26 week follow-up, and 52 week follow-up
Quality of Life Inventory (QOLI) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in QOLI at post-treatment, 26 week follow-up, and 52 week follow-up
EuroQol-5 dimension (EQ5D) | Baseline, post-treatment (variable depending on disorder), 26 feel follow-up, 52 week follow-up
  Change in EQ5D at post-treatment, 26 week follow-up, and 52 week follow-up
Sheehan Disability Scales (SDS) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in SDS at post-treatment, 26 week follow-up, and 52 week follow-up
Self-rated health 5 (SRH-5) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in SRH-5 at post-treatment, 26 week follow-up and 52 week follow-up
Obsessive Compulsive Inventory-Revised (OCI-R) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in OCI-R at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Liebowitz Social Anxiety Scale Self-report (LSAS-SR) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in LSAS-SR at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Panic Disorder Severity Scale Self-rated (PDSS-SR) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in PDSS-SR at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Penn-State Worry Questionnaire (PSWQ) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in PSWQ at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Post Traumatic Stress Disorder Symptom Scale-Self report (PTSDSS) | Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
  Change in PTSDSS at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.

OTHER OUTCOMES:
Inflammatory cytokines | Baseline, post-treatment (variable depending on disorder)
  Change in inflammatory cytokines at post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet and Gustavsberg primary care center, Stockholm, Stockholm County, Sweden